CLINICAL TRIAL: NCT04435392
Title: A Phase I/II Study Of The Efficacy,Safety and PharmacokineticsOf Jaktinib Hydrochloride Cream In Subjects With Mild To Moderate Atopic Dermatitis
Brief Title: Jaktinib Hydrochloride Cream For Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAKT002
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Jaktinib
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: Cohort 1, 0.5% Jaktinib Bid (Experimental): Subjects were randomly assigned to receive either Jaktinib cream or a placebo in a ratio of 3 to 1.The Jaktinib hydrochloride 0.5% Cream will be applied topically twice daily.
  Interventions: Drug: Jaktinib Hydrochloride Cream; Drug: Placebo
- Part 1: Cohort 2,1.5% Jaktinib Bid (Experimental): Subjects were randomly assigned to receive either Jaktinib cream or a placebo in a ratio of 3 to 1.The Jaktinib hydrochloride 1.5% Cream will be applied topically twice daily.
  Interventions: Drug: Jaktinib Hydrochloride Cream; Drug: Placebo
- Part 1: Cohort 3, 2.5% Jaktinib Qd (Experimental): Subjects were randomly assigned to receive either Jaktinib cream or a placebo in a ratio of 3 to 1.The Jaktinib hydrochloride 2.5% Cream will be applied topically Once daily.
  Interventions: Drug: Jaktinib Hydrochloride Cream; Drug: Placebo
- Part 1: Cohort 4, 2.5% Jaktinib Bid (Experimental): Subjects were randomly assigned to receive either Jaktinib cream or a placebo in a ratio of 3 to 1.The Jaktinib hydrochloride 2.5% Cream will be applied topically twice daily.
  Interventions: Drug: Jaktinib Hydrochloride Cream; Drug: Placebo
- Dose extension: Vehicle Control (Placebo Comparator): the Vehicle Control cream will be applied topically twice daily
  Interventions: Drug: Placebo
- Dose extension: low-dose group, X% (Experimental): X% based on results of part 1. The Jaktinib Hydrochloride X% Cream will be applied topically twice daily
  Interventions: Drug: Jaktinib Hydrochloride Cream
- Dose extension: high-dose group, Y% (Experimental): Y% based on results of part 1. The Jaktinib Hydrochloride Y% Cream will be applied topically twice daily
  Interventions: Drug: Jaktinib Hydrochloride Cream

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Cream — Subjects in each group were scheduled to give the drug for 8 weeks.
  Other Names: Jaktinib
  Arms: Dose extension: high-dose group, Y%; Dose extension: low-dose group, X%; Part 1: Cohort 1, 0.5% Jaktinib Bid; Part 1: Cohort 2,1.5% Jaktinib Bid; Part 1: Cohort 3, 2.5% Jaktinib Qd; Part 1: Cohort 4, 2.5% Jaktinib Bid
Drug: Placebo — Placebo
  Arms: Dose extension: Vehicle Control; Part 1: Cohort 1, 0.5% Jaktinib Bid; Part 1: Cohort 2,1.5% Jaktinib Bid; Part 1: Cohort 3, 2.5% Jaktinib Qd; Part 1: Cohort 4, 2.5% Jaktinib Bid

SUMMARY:
This study includes a dose escalation part and a dose extension part.

DETAILED DESCRIPTION:
In the dose-increasing part, a multicenter, dose-increasing, randomized, double-blind, placebo-parallel control design was adopted. Subjects were enrolled into different dose groups in sequence according to the inclusion sequence, and each group was scheduled to give the drug for 8 weeks.Subjects in each group were observed for 4 weeks after administration. When the number of ≥2 grade drug-related adverse events (cases) was less than 50%, subjects in the next group could be enrolled.Otherwise, IDMC will decide whether to continue the next set of tests.Subjects in each group were randomly assigned to receive either Jaktinib cream (6 cases) or placebo (2 cases) in a ratio of 3 to 1.A total of 32 subjects are expected to be enrolled in 6 centers.

The dose expansion was a multicenter, randomized, double-blind, placebo-parallel control design in which subjects were randomly assigned to 3 groups (1 placebo group and 2 experimental drugs group).It is estimated that a total of 60 subjects will be enrolled in about 15 centers. This part is divided into two stages.Stage 2 test (9 ~ 16 weeks) : Extension test.

ELIGIBILITY:
Inclusion Criteria:

* 18~ 65 years old (including boundary value), gender is not limited;
* Have a clinical diagnosis of atopic dermatitis;
* Have a PGA(Physician's Global Assessment) score of 2 (mild) or 3 (moderate) at baseline;
* The total area of atopic dermatitis is about 10%~20% of the total area of the body surface at baseline.

Exclusion Criteria:

* Evidence of certain skin conditions/infections at baseline;
* Have certain laboratory abnormalities at baseline;
* Females who are pregnant, breastfeeding, or are of childbearing potential not using highly effective contraception;
* Other conditions that the investigators considered inappropriate to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Physician's Global Assessment (PGA) Response of Clear or Almost Clear | 7 days after the last dose
  A total PGA score of 0 or 1 or a decrease of ≥2 from baseline

SECONDARY OUTCOMES:
Proportion of Participants With Response of Clear or Almost Clear From Baseline | Treatment at 8,16 weeks
  PGA score of 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, PhD, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China